CLINICAL TRIAL: NCT02388568
Title: A Randomized Controlled Trial of Lifestyle Modification and Lorcaserin for Weight Loss Maintenance
Brief Title: Lifestyle Modification and Lorcaserin for Weight Loss Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eisai-819111
Record Dates: First submitted 2015-01-29; First posted 2015-03-17 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lorcaserin plus Lifestyle Modification (Active Comparator)
  Interventions: Drug: Lorcaserin
- Placebo plus Lifestyle Modification (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorcaserin — Lorcaserin plus Lifestyle Modification
  Arms: Lorcaserin plus Lifestyle Modification
Drug: Placebo — Placebo plus Lifestyle Modification
  Arms: Placebo plus Lifestyle Modification

SUMMARY:
The proposed 12-month randomized controlled trial will assess the efficacy of lifestyle counseling, combined with lorcaserin (10 mg BID) or placebo, in maintaining weight loss achieved during a prior 14-week dietary run-in.

14-week run-in. To qualify for randomization, participants must lose ≥5% of initial weight in the 14-week dietary run-in. This loss will be achieved with the provision of weekly, group lifestyle counseling, which includes a 1000-1200 kcal/day portion-controlled diet that combines four daily servings of a liquid diet (HMR shakes) with an evening meal of a frozen-food entree (and a fruit and vegetable serving). More than 70% of participants are expected to achieve the 5% criterion loss during the 14-week run-in.

A total of 182 women and men with a BMI ≥33 and ≤55 kg/m2, without co-morbidities, or ≥30 and ≤55 kg/m2 (with a co-morbid cardiovascular disease (CVD) condition) will be enrolled in the 4-month run-in period. Prior to enrollment, all participants will have a history, physical exam, electrocardiogram (EKG), and appropriate blood tests. They will attend weekly group sessions for 14 weeks. Participants will have a brief medical visit at week 8 to check their health and blood tests will be repeated. The investigators anticipate that 136 (75%) participants will lose 5% or more of initial weight and qualify for randomization. Participants who do not lose 5% will be provided a list of weight loss resources (e.g., other programs) to facilitate their continued weight management.

12-month randomized trial with lorcaserin. A total of 136 participants who have lost 5% or more of initial weight in the run-in period will be randomly assigned, in double-blind fashion, to lorcaserin (10 mg BID) or matching placebo. To be eligible, participants must have a BMI (after prior weight loss) ≥30 kg/m2 (without co-morbidities) or greater than or equal to ≥27 (with a co-morbidity). Randomization will be performed by the Investigational Drug Service at the Hospital of the University of Pennsylvania. Prior to randomization, all participants will complete a second brief history and physical examination, as well as an EKG and blood tests. Medication will be dispensed at the randomization visit and at brief medical visits that follow. Over the 1 year, all participants will participate in 16 group lifestyle modification classes designed for weight loss maintenance, approximately half of which will be delivered by group conference call.

Primary outcome measure. The primary endpoint is change in body weight (in kg), as measured from randomization to month 12. The co-primary end-point is the percentage of participants in the two groups that, at month 12, maintained the ≥5% reduction in body weight achieved during the 14-week dietary run-in period. Secondary efficacy endpoints include changes in CVD risk factors, glycemic control, and quality of life, as measured from randomization to month 12. Exploratory endpoints include changes in these CVD and related outcomes, as measured at the start of the 14-week run-in period to month 12. The investigators also will examine the percentage of participants in the two groups who at month 12 achieved losses of ≥5%, ≥10%, and ≥15% of initial weight, as measured from the start of the run-in period.

Safety endpoints will include physical examination, electrocardiogram, adverse events (AEs), standard laboratory tests, and mental health assessed by the Columbia Suicidality Severity Rating Scale (C-SSRS) and Patient Health Questionnaire (PHQ-9).

Statistical Analysis. The planned sample size of 136 participants, with a 1:1 randomization ratio, assumes a 20% drop-out rate (at month 12) and was estimated to be adequate to evaluate the primary endpoint with power ≥90% (P=0.05, two-sided test). The investigators predict a difference in weight change between the two groups (from randomization to month 12) of 4 kg (SD=3.5). Pre-specified data analysis will be performed on the full analysis set, comprising all randomized individuals exposed to trial drug with at least one post-randomization weight assessment.

ELIGIBILITY:
Inclusion Criteria (for the Randomized Controlled Trial)

1. Participants must have lost ≥ 5% of initial weight in the group lifestyle modification program (during the 14-week diet run-in period).
2. Participants must have a BMI ≥ 30 and ≤ 55 kg/m² or have a BMI ≥ 27 kg/m² with a obesity-related co-morbid condition
3. Age ≥ 21 years and ≤ 65
4. Eligible female patients will be:

   * non-pregnant, evidenced by a negative urine dipstick pregnancy test
   * non-lactating
   * surgically sterile or postmenopausal, or they will agree to continue to use an accepted method of birth control during the study
5. Participants must have a primary care provider (PCP) who is responsible for providing routine care and have a reliable telephone service with which to participate in conference calls

Exclusion Criteria:

1. Pregnant or nursing (or plans to become pregnant in the next 18 months)
2. Current major depressive episode, active suicidal ideation, or history of suicide attempts
3. Use in the past 14 days of monoamine oxidase inhibitors, selective serotonin reuptake inhibitors (SSRI), serotonin-norepinephrine reuptake inhibitors (SNRI), tricyclics, lithium, triptans, antipsychotics, cabergoline, linezolid, tramadol, dextromethorphan, tryptophan, bupropion, St. John's Wort, or medicines to treat erectile dysfunction
4. Uncontrolled hypertension (systolic blood pressure ≥ 160 mm Hg, or diastolic blood pressure ≥ 100 mm Hg)
5. Type 1 diabetes or type 2 diabetes
6. A fasting glucose ≥ 126 mg/dl or HbA1c ≥ 6.5
7. Recent history of cardiovascular disease (e.g., myocardial infarction or stroke within the past 6 months), congestive heart failure, or heart block greater than first degree
8. Clinically significant hepatic or renal disease
9. Thyroid disease not controlled
10. History of malignancy (except for non-melanoma skin cancer)
11. Use of medications known to induce significant weight loss/gain, including chronic use of oral steroids
12. Psychiatric hospitalization within the past 6 months
13. Self-reported alcohol or substance abuse within the past 12 months, including at-risk drinking (current consumption of ≥ 14 alcoholic drinks per week)
14. Loss of ≥ 10 lb of body weight within the past 3 months
15. History of (or plans for) bariatric surgery

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Wadden, Ph.D., Principal Investigator — University of Pennsylvania; Robert I Berkowitz, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Pearl RL, Wadden TA, Chao AM, Walsh O, Alamuddin N, Berkowitz RI, Tronieri JS. Weight Bias Internalization and Long-Term Weight Loss in Patients With Obesity. Ann Behav Med. 2019 Jul 17;53(8):782-787. doi: 10.1093/abm/kay084. PMID 30304382
- [Derived] Pearl RL, Wadden TA, Allison KC, Chao AM, Alamuddin N, Berkowitz RI, Walsh O, Tronieri JS. Causal Attributions for Obesity Among Patients Seeking Surgical Versus Behavioral/Pharmacological Weight Loss Treatment. Obes Surg. 2018 Nov;28(11):3724-3728. doi: 10.1007/s11695-018-3490-7. PMID 30191502
- [Derived] Pearl RL, Wadden TA, Tronieri JS, Berkowitz RI, Chao AM, Alamuddin N, Leonard SM, Carvajal R, Bakizada ZM, Pinkasavage E, Gruber KA, Walsh OA, Alfaris N. Short- and Long-Term Changes in Health-Related Quality of Life with Weight Loss: Results from a Randomized Controlled Trial. Obesity (Silver Spring). 2018 Jun;26(6):985-991. doi: 10.1002/oby.22187. Epub 2018 Apr 20. PMID 29676530
- [Derived] Shaw Tronieri J, Wadden TA, Berkowitz RI, Chao AM, Pearl RL, Alamuddin N, Leonard SM, Carvajal R, Bakizada ZM, Pinkasavage E, Gruber KA, Walsh OA, Alfaris N. A Randomized Trial of Lorcaserin and Lifestyle Counseling for Maintaining Weight Loss Achieved with a Low-Calorie Diet. Obesity (Silver Spring). 2018 Feb;26(2):299-309. doi: 10.1002/oby.22081. Epub 2017 Dec 29. PMID 29288545
- [Derived] Tronieri JS, Alfaris N, Chao AM, Pearl RL, Alamuddin N, Bakizada ZM, Berkowitz RI, Wadden TA. Lorcaserin plus lifestyle modification for weight loss maintenance: Rationale and design for a randomized controlled trial. Contemp Clin Trials. 2017 Aug;59:105-112. doi: 10.1016/j.cct.2017.06.004. Epub 2017 Jun 16. PMID 28600158
- [Derived] Pearl RL, Wadden TA, Hopkins CM, Shaw JA, Hayes MR, Bakizada ZM, Alfaris N, Chao AM, Pinkasavage E, Berkowitz RI, Alamuddin N. Association between weight bias internalization and metabolic syndrome among treatment-seeking individuals with obesity. Obesity (Silver Spring). 2017 Feb;25(2):317-322. doi: 10.1002/oby.21716. PMID 28124502

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lorcaserin Plus Lifestyle Modification | Placebo Plus Lifestyle Modification
Started | 69 | 68
Completed | 59 | 53
Not Completed | 10 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lorcaserin Plus Lifestyle Modification | Placebo Plus Lifestyle Modification | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (10.5) | 47.7 (9.8) | 46.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 59 | 118
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 49 | 45 | 94
  White | 15 | 18 | 33
  Asian | 2 | 2 | 4
  Multiracial or other | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 4 | 3 | 7
Height [Mean (Standard Deviation); unit: cm] | 168.8 (8.6) | 165.7 (9.4) | 167.2 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight (kg)
Description: This is the change in weight from randomization to week 52. This does not include the weight loss in the 14-week LCD.
Time Frame: 52 weeks post-randomization
Measure: Mean (Standard Error); unit: kg
Arm/Group | Lorcaserin Plus Lifestyle Modification | Placebo Plus Lifestyle Modification
Number analyzed (Participants) | 69 | 68
kg | 2.0 (0.8) | 2.5 (0.8)

2. Primary Outcome: Proportion Maintaining >= 5% Loss of Initial Weight
Description: This is the number of participants who maintained >=5% loss of initial weight in the randomization to week 52 trial period.
Time Frame: 52 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Lorcaserin Plus Lifestyle Modification | Placebo Plus Lifestyle Modification
Number analyzed (Participants) | 69 | 68
Participants | 38 | 29

3. Secondary Outcome: Body Weight (% Change)
Description: The % change in body weight from randomization to week 52.
Time Frame: 52 weeks post-randomization
Measure: Mean (Standard Error); unit: % change
Arm/Group | Lorcaserin Plus Lifestyle Modification | Placebo Plus Lifestyle Modification
Number analyzed (Participants) | 69 | 68
% change | 1.8 (0.8) | 2.2 (0.8)

4. Secondary Outcome: Proportion Maintaining >= 10% Loss of Initial Weight
Description: This is the number of participants who maintained >=10% loss of initial weight in the randomization to week 52 trial period.
Time Frame: 52 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Lorcaserin Plus Lifestyle Modification | Placebo Plus Lifestyle Modification
Number analyzed (Participants) | 69 | 68
Participants | 20 | 20

5. Secondary Outcome: Body Weight
Description: This is the change in weight from baseline (screening visit) to the final week 52 medical assessment visit.
Time Frame: -14 week (start of LCD program) to week 52
Measure: Mean (Standard Error); unit: kg
Arm/Group | Lorcaserin Plus Lifestyle Modification | Placebo Plus Lifestyle Modification
Number analyzed (Participants) | 69 | 68
kg | -9.4 (0.9) | -7.5 (1.0)

6. Secondary Outcome: Body Weight (% Change)
Description: This is the change in weight from the baseline (screening visit) to the final week 52 medical assessment visit.
Time Frame: -14 week (start of LCD program) to week 52
Measure: Mean (Standard Error); unit: % change
Arm/Group | Lorcaserin Plus Lifestyle Modification | Placebo Plus Lifestyle Modification
Number analyzed (Participants) | 69 | 68
% change | -7.8 (0.8) | -6.6 (0.9)

ADVERSE EVENTS:
Time Frame: Adverse events for phase 2 of the trial were reported from the time of randomization to 13 months after randomization. Safety assessments included recording adverse events at all clinic visits; a physical examination, fasting blood test, and urine pregnancy test (as appropriate) at randomization, and weeks 24 and 52 of phase 2; and nine brief medical visits to measure vital signs, review health, and administer the Columbia-Suicide Severity Rating Scale.
Arm/Group | Lorcaserin Plus Lifestyle Modification | Placebo Plus Lifestyle Modification
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/68
Serious Adverse Events (participants affected / at risk) | 2/69 | 8/68
Other Adverse Events (participants affected / at risk) | 56/69 | 49/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorcaserin Plus Lifestyle Modification (N=69) | Placebo Plus Lifestyle Modification (N=68)
Sialolithiasis/sialadenitis (Endocrine disorders) | 1 | 0
Staph cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cholelithiasis (Gastrointestinal disorders) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1
Lung nodules (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pregnancy (Reproductive system and breast disorders) | 0 | 1
Vertigo (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lorcaserin Plus Lifestyle Modification (N=69) | Placebo Plus Lifestyle Modification (N=68)
Headache (Nervous system disorders) | 12 | 7
Fatigue (General disorders) | 11 | 12
Constipation (Gastrointestinal disorders) | 10 | 3
Dry mouth (General disorders) | 7 | 3
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Dizziness (General disorders) | 4 | 2
Musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-01-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT02388568/Prot_000.pdf
  • Statistical Analysis Plan (2014-02-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT02388568/SAP_001.pdf